CLINICAL TRIAL: NCT06542497
Title: Randomized, Double-masked, Placebo-controlled, Multicenter Study of the Efficacy and Safety of Phentolamine Ophthalmic Solution (POS) 0.75% in Participants With Presbyopia
Brief Title: Evaluate Efficacy and Safety of POS to Improve Distance-corrected Near Visual in Participants With Presbyopia
Acronym: VEGA-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPI-NYXP-302
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-masked, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.75% phentolamine ophthalmic solution (Active Comparator): Drug: phentolamine ophthalmic solution 0.75%, a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Interventions: Drug: 0.75% phentolamine ophthalmic solution
- phentolamine ophthalmic solution vehicle (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.75% phentolamine ophthalmic solution — Once daily dosing
  Other Names: Nyxol
  Arms: 0.75% phentolamine ophthalmic solution
Drug: Placebo — Once daily dosing
  Other Names: phentolamine ophthalmic solution vehicle
  Arms: phentolamine ophthalmic solution vehicle

SUMMARY:
Safety and efficacy of POS in participants with presbyopia

DETAILED DESCRIPTION:
Randomized, Double-Masked, Placebo-Controlled, Multicenter, Phase 3 Study of the Efficacy and Safety of Phentolamine Ophthalmic Solution (POS) 0.75% in Participants with Presbyopia

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Males or females ≥ 45 and ≤ 64 years of age
2. Able to comply with all protocol-mandated procedures independently and to attend all scheduled office visits
3. Able and willing to give signed informed consent
4. Able to self-administer study medication throughout the study period

   Inclusion criteria #5, #6, and #7 must all be met at both Screening and Baseline Visits:
5. BCDVA of 55 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (20/20 Snellen equivalent) or better in photopic conditions in each eye
6. DCNVA of 50 ETDRS letters (20/50 Snellen equivalent) or worse but not <35 ETDRS letters (20/100 Snellen equivalent) in photopic conditions in each eye and binocularly
7. For participants who depend on reading glasses or bifocals, binocular best-corrected near VA of 65 ETDRS letters (20/25 Snellen equivalent) or better
8. Photopic PD of ≥ 4 mm in the study eye at Screening

Exclusion Criteria:

Excluded from the study will be individuals with any of the following characteristics:

Ophthalmic (in either eye):

1. Use of any topical prescription (including Vuity® or Qlosi™) or over-the-counter (OTC) ophthalmic medications of any kind within 7 days of Screening until study completion, with the exception of lid scrubs with OTC products (eg, OCuSOFT® lid scrub, SteriLid®, baby shampoo, etc.) and artificial tears as specified in Exclusion Criterion #2 below
2. Use of any OTC artificial tears (preserved or unpreserved) during visit days or 15 min before or after instillation of study medication
3. Use of Ryzumvi™ (POS) within 7 days prior to Screening
4. Use of any dry eye product, such as topical ophthalmic therapy for dry eye (eg, generic cyclosporine, Restasis®, Xiidra®, Cequa®, Eysuvis®, and Meibo®) or intranasal dry eye product (eg, Tyrvaya®) or other devices within 12 months prior to Screening
5. Tear break-up time of < 5 seconds or corneal fluorescein staining (CFS) Grade ≥ 2 in the inferior zone or Grade ≥ 1 in the central zone using the National Eye Institute scale
6. Clinically significant ocular disease (eg, cataract, glaucoma, corneal edema, uveitis, retinal degeneration, loss of visual field, or any macular pathology) that, in the judgment of the Investigator, might interfere with study procedures
7. Recent or current evidence of ocular infection or inflammation in either eye (such as current evidence of clinically significant blepharitis, conjunctivitis, keratitis, etc.). Participants must be symptom free for at least 7 days prior to Screening
8. Any history of herpes simplex or herpes zoster keratitis
9. Known allergy, hypersensitivity, or contraindication to any component of the phentolamine or vehicle formulations
10. Prior participation in a study involving the use of POS for the treatment of presbyopia or night vision disturbance
11. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal
12. Ocular trauma within 6 months prior to Screening
13. Ocular surgery or any ocular laser treatment within 6 months prior to Screening. Any history of radial keratotomy is prohibited
14. Participants with surgical monovision, multifocal, or extended depth-of-focus intraocular lenses (IOLs). Monofocal IOLs are acceptable if in place > 6 months prior to Screening
15. Monofocal IOL in place > 6 months prior to Screening with any posterior capsule opacification
16. History of any traumatic (surgical or nonsurgical) or nontraumatic condition affecting the pupil or iris (eg, irregularly shaped pupil, neurogenic pupil disorder, iris atrophy, iridotomy, iridectomy, iritis, etc.)
17. Unwilling or unable to discontinue use of contact lenses at least 1 hour prior to Screening for soft contact lenses or at least 8 hours prior to Screening for hard gas permeable contact lenses, and at least 8 hours (for both types of lenses) prior to all other office visits

    Systemic:
18. Known hypersensitivity or contraindication to alpha- and/or beta-adrenoceptor antagonists (eg, chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure (BP) or heart rate (HR); second- or third-degree heart blockage or congestive heart failure)
19. Known hypersensitivity or contraindication to any systemic cholinergic parasympathomimetic agent
20. Clinically significant systemic disease (eg, uncontrolled diabetes, myasthenia gravis, cancer, hepatic, renal, endocrine, or cardiovascular disorders) that might interfere with the study as deemed by the judgment of the Investigator
21. Initiation of treatment with, or any changes to, the current dosage, drug, or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to Screening or during the study; however, Flomax® (tamsulosin) is specifically excluded
22. Participation in any investigational study within 30 days prior to Screening
23. Females of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. Acceptable methods include the use of at least one of the following: intrauterine device, hormonal contraception (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence. A female is considered to be of childbearing potential unless she is 1 year postmenopausal or 3 months post-surgical sterilization. All females of childbearing potential, including those with post-tubal ligation, must have a negative urine pregnancy test result at Visit 1 (Screening)
24. Resting HR outside the range of 50 to 110 beats per min (bpm) following at least a 5 min rest period in the sitting position at Visit 1 (Screening). HR may be repeated only once if outside the specified range, following another 5 min rest period in the sitting position
25. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg following at least a 5-min rest period in the sitting position at Visit 1 (Screening). BP may be repeated only once if outside the specified range, following another 5-min rest period in the sitting position

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 545 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | Day 8
  The primary efficacy endpoint is the percentage of participants with ≥ 15 letters of improvement in binocular DCNVA and with < 5 letters of loss in binocular BCDVA from baseline comparing POS-treated participants to placebo-treated participants at 12 hours post-dose at Visit 4 (Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Jay V Pepose, MD, Study Chair — Ocuphire Pharma
Locations (13):
- United States (13):
  - United States, Phoenix, Arizona
  - United States, Scottsdale, Arizona
  - United States, Glendale, California
  - United States, Newport Beach, California
  - United States, Delray Beach, Florida
  - United States, Longwood, Florida
  - United States, Rochester, New York
  - United States, Garner, North Carolina
  - United States, Athens, Ohio
  - United States, Warwick, Rhode Island
  - United States, Goodlettsville, Tennessee
  - United States, Memphis, Tennessee
  - United States, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No